CLINICAL TRIAL: NCT05261672
Title: Midazolam as an Adjuvant to Bupivacaine in Quadratus Lumborum Block After Caesarean Section; Does it Offer Better Pain Control? a Randomized Double Blind Clinical Trial
Brief Title: Regional Midazolam in Quadratus Lumborum Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, prof., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB022022
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain
Keywords: Midazolam; Bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Midazolam; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group QL1 (Active Comparator): quadratus lumborum block will be done. 20 ml bupivacaine 0.25% will be injected + 1 ml saline on each side
  Interventions: Drug: Bupivacain
- Group QL2 (Active Comparator): quadratus lumborum block will be done. ) 20 ml bupivacaine 0.25% will be injected + 2 mg midazolam in 1 ml saline on each side.
  Interventions: Drug: Midazolam/ bupivaciane

INTERVENTIONS:
Drug: Midazolam/ bupivaciane — 20 ml bupivacaine 0.25% will be injected + 2 mg midazolam in 1 ml saline on each side.
  Arms: Group QL2
Drug: Bupivacain — 20 ml bupivacaine 0.25% will be injected + 1 ml saline on each side
  Arms: Group QL1

SUMMARY:
Midazolam has been used in regional anesthesia of brachial plexus block; it has offered accepted postoperative pain relief. This study will use it in as an adjuvant to bupivacaine 0.25% in quadratus lumborum block in caesarean section

DETAILED DESCRIPTION:
It is vital to apply adequate postoperative analgesia following Caesarean section (C-section), since it will affect the distinct surgical recovery requirements of the parturient. The ultrasound-guided quadratus lumborum block (QLB), first introduced by Blanco R. in 2007, has been recognized as an effective abdominal wall block approach, in which local anesthetic injected from the posterior abdomen will spread around the quadratus lumborum muscle and block the intermuscular nerves. In addition, such block is also closely related to multiple sympathetic fibres and is connected to the thoracic paravertebral space. Typically, QLB is found to be effective, which can provide satisfactory analgesic effect.

Midazolam is one of the clinically water-soluble benzodiazepines and effective to produce the analgesic effect through the neuraxial pathways. The organs and joints of humans have the benzodiazepine receptor, and midazolam is revealed to produce the analgesic effect through the gamma-aminobutyric acid receptors (GABA) in the spinal cord. Previous studies have reported that the midazolam (75 μg/kg) through the intraarticular route can decrease the pain intensity for arthroscopic knee surgery. In addition, the intrathecal midazolam (2 mg) is reported to prolong the duration of analgesia without any adverse effects following knee arthroscopies. Perineural midazolam has been also evaluated in brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* age from 24 to 40 years old
* weight from 50 to 80 kg,
* normal singleton pregnancy with a gestation of at least 37 weeks

Exclusion Criteria:

* Coagulopathy
* maternal anatomic abnormalities in the block region
* localized infection
* incapable of comprehending or using the verbal rating pain scoring system
* Included medications allergy
* history of chronic pain or regular opioid use.

Ages: 24 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy with a gestation of at least 37 weeks
Enrollment: 60 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
rescue analgesia | 24 hours
  Time to rescue analgesia in the post operative period

SECONDARY OUTCOMES:
Visual analog scale | 2, 4, 6, 8, 12, 16, 20, 24 hours
  Pain Visual analog scale during the 1st 24 hours

OTHER OUTCOMES:
total Analgesic requirement | first 24 hours
  total Analgesic requirement in the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Ishio J, Komasawa N, Kido H, Minami T. Evaluation of ultrasound-guided posterior quadratus lumborum block for postoperative analgesia after laparoscopic gynecologic surgery. J Clin Anesth. 2017 Sep;41:1-4. doi: 10.1016/j.jclinane.2017.05.015. Epub 2017 Jun 1. PMID 28802593
- [Result] Tucker AP, Mezzatesta J, Nadeson R, Goodchild CS. Intrathecal midazolam II: combination with intrathecal fentanyl for labor pain. Anesth Analg. 2004 Jun;98(6):1521-1527. doi: 10.1213/01.ANE.0000112434.68702.E4. PMID 15155300
- [Result] Lefevre N, Klouche S, de Pamphilis O, Herman S, Gerometta A, Bohu Y. Peri-articular local infiltration analgesia versus femoral nerve block for postoperative pain control following anterior cruciate ligament reconstruction: Prospective, comparative, non-inferiority study. Orthop Traumatol Surg Res. 2016 Nov;102(7):873-877. doi: 10.1016/j.otsr.2016.07.011. Epub 2016 Oct 4. PMID 27720193